CLINICAL TRIAL: NCT07138885
Title: A Phase II, Single-Arm, Prospective Trial on the Efficacy and Safety of QL1706 Combination Regimen as Second-Line Therapy for Targeted-Immunotherapy-Resistant Hepatocellular Carcinoma
Acronym: DRIVE-II
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Tian-Qi Zhang, Associate Professor, Associate Chief Physician, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRIVE-II
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma (HCC); Second Line Treatment
Keywords: Second line treatment; Hepatocellular Carcinoma (HCC); Immunotherapy resistance
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Bevacizumab; trifluridine tipiracil drug combination

STUDY DESIGN:
Intervention Model Description: Arm 1: To evaluate the objective response rate (ORR) of HAI-FOLFOX + bevacizumab + QL1706 in patients with intermediate-advanced hepatocellular carcinoma (HCC) who developed resistance or recurrence after prior treatment with surgical resection/ablation/TACE combined with TKIs and/or PD-(L)1 inhibitors.
  Arm 2: To evaluate the objective response rate (ORR) of TACE + bevacizumab + TAS-102 + QL1706 in patients with intermediate-advanced HCC who developed resistance or recurrence after prior HAI-FOLFOX combined with TKIs and/or PD-(L)1 inhibitors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAI-FOLFOX + bevacizumab + QL1706 (Experimental): To evaluate the objective response rate (ORR) of HAI-FOLFOX + bevacizumab + QL1706 in patients with intermediate-advanced hepatocellular carcinoma (HCC) who developed resistance or recurrence after prior treatment with surgical resection/ablation/TACE combined with TKIs and/or PD-(L)1 inhibitors.
  Interventions: Procedure: HAI-FOLFOX + bevacizumab + QL1706
- TACE + bevacizumab + QL1706 + TAS-102 (Experimental): To evaluate the objective response rate (ORR) of TACE + bevacizumab + TAS-102 + QL1706 in patients with intermediate-advanced HCC who developed resistance or recurrence after prior HAI-FOLFOX combined with TKIs and/or PD-(L)1 inhibitors.
  Interventions: Procedure: TACE + bevacizumab + TAS-102 + QL1706

INTERVENTIONS:
Procedure: HAI-FOLFOX + bevacizumab + QL1706 — Arm 1:
  HAI-FOLFOX Administration (Day 1 of Each Cycle) Super-selective insertion the arterial catheter into the tumor-feeding artery, then infusion: Oxaliplatin: 85 mg/m², Leucovorin: 400 mg/m², 5-FU: 2500 mg/m²
  Administer bevacizumab (7.5 mg/kg; total dose capped at 300 mg or 400 mg) via arterial infusion.
  Then QL1706 (5 mg/kg, IV infusion, Q3W).
  Treatment Schedule: Repeat HAI-FOLFOX + arterial bevacizumab every 3 weeks (max 6 cycles), followed by QL1706 maintenance (Q3W).
  Other Names: HAI-FOLFOX; bevacizumab; QL1706
  Arms: HAI-FOLFOX + bevacizumab + QL1706
Procedure: TACE + bevacizumab + TAS-102 + QL1706 — Arm 2:
  On-Demand TACE (Lipiodol: ≤10 mL, mixed with platinum + doxorubicin agent, each ≤50 mg) to form an emulsion. Repeat TACE until TACE resistance develops (typically ~4 sessions).
  Administer bevacizumab (7.5 mg/kg; total dose capped at 300 mg or 400 mg) via intra-arterial route.
  After first TACE, begin TAS-102 (15 mg/m² po BID) once liver function recovers to acceptable levels.
  Then QL1706 (5 mg/kg, IV infusion, Q3W).
  Other Names: bevacizumab; TAS-102; QL1706; TACE
  Arms: TACE + bevacizumab + QL1706 + TAS-102

SUMMARY:
The goal of this prospective Phase II clinical trial is to evaluate the efficacy and safety of QL1706-based combination therapy in patients with hepatocellular carcinoma (HCC) who have failed prior targeted-immunotherapy (e.g., anti-PD-1/PD-L1 + antiangiogenic therapy).

The main question is:

Can the combination of localized-regional therapy (e.g., HAIC/TACE) and systemic dual immunotherapy (QL1706) overcome resistance and improve outcomes in second-line HCC treatment?

Participants will:

1. Receive QL1706 (a dual immune checkpoint inhibitor) combined with either:

   Hepatic arterial infusion chemotherapy (HAIC)/transarterial chemoembolization (TACE), or Antiangiogenic targeted therapy.
2. Undergo regular imaging (e.g., MRI/CT) and biomarker assessments for efficacy monitoring.
3. Be evaluated for adverse events (AEs) and quality of life.

This study seeks to establish a novel therapeutic paradigm for HCC patients after targeted-immunotherapy failure, addressing the unmet need for evidence-based second-line strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary Participation, Willingly signs the written informed consent form.
2. Aged 18-65 years (inclusive), any gender.
3. Histologically, cytologically, or clinically confirmed hepatocellular carcinoma (HCC) with disease progression after first-line targeted therapy combined with immunotherapy, or intolerable to first-line targeted-immunotherapy combination treatment.
4. No prior exposure to VEGF monoclonal antibodies, CTLA-4 inhibitors, or bispecific antibodies. For arm 1: No prior treatment with oxaliplatin or fluorouracil-based drugs.
5. Liver Function: Child-Pugh class A or class B (score ≤7), with no history of hepatic encephalopathy.
6. Performance Status: ECOG PS score 0 or 1.
7. Life Expectancy ≥12 weeks.
8. Measurable Lesion: ≥1 measurable target lesion per RECIST v1.1 (not previously irradiated/localized; lesions in prior treatment areas are acceptable if progression is confirmed).
9. Preserved organ & bone marrow function (within 7 days before treatment; no blood products/growth factors within 14 days prior):

   * Neutrophil count (ANC) ≥1.5×10⁹/L
   * Platelets ≥75×10⁹/L
   * Hemoglobin ≥90 g/L
   * Albumin ≥28 g/L
   * ALT/AST/Alkaline phosphatase (AKP) ≤3×ULN
   * Total bilirubin (TBIL) ≤2×ULN
   * INR ≤2 or PT prolongation ≤6 sec above ULN
   * Urine protein <2+ (if ≥2+, 24-hour urine protein must be <1.0 g).
10. Viral Hepatitis Management

    * If HBsAg-positive: HBV DNA <2000 IU/mL or 10⁴ copies/mL, with ongoing antiviral therapy (entecavir/tenofovir disoproxil fumarate/tenofovir alafenamide/emtecavir).
    * HCV-infected patients with undetectable HCV RNA are considered HCV-negative.
11. Contraception

    * Fertile participants (male/female) must use reliable contraception (hormonal/barrier/abstinence) during and for ≥180 days post-treatment.
    * Women of childbearing potential must have a negative serum pregnancy test within 7 days before enrollment.

Exclusion Criteria:

1. Histologically/cytologically confirmed fibrolamellar HCC, sarcomatoid HCC, cholangiocarcinoma, or mixed hepatocellular-cholangiocarcinoma.
2. Other active malignancies within 5 years prior to enrollment, except cured localized tumors (e.g., basal cell carcinoma, squamous cell skin cancer, superficial bladder cancer, in situ prostate/cervical/breast cancer).
3. History of or planned liver transplantation.
4. Clinically significant ascites requiring therapeutic paracentesis, uncontrolled pleural/pericardial effusion (asymptomatic minimal ascites on imaging allowed).
5. Known CNS metastases or leptomeningeal disease.
6. Tumor thrombus involving both main portal vein and superior mesenteric vein, or portal vein and inferior vena cava.
7. High-risk variceal bleeding:

   * Esophageal/gastric variceal bleeding within 6 months
   * High-grade varices on endoscopy within 3 months
   * Portal hypertension with bleeding risk (splenomegaly, active ulcers, occult blood+, or endoscopic "red signs").
8. Life-threatening hemorrhage within 3 months requiring transfusion/surgery/medical intervention.
9. Significant bleeding risk:

   * Hemoptysis/tumor bleeding within 2 weeks
   * Thromboembolism within 6 months
   * Therapeutic anticoagulation (except prophylactic LMWH) within 2 weeks
   * Antiplatelet therapy (aspirin >325 mg/day, clopidogrel >75 mg/day) within 10 days
   * Tumor invasion of major vessels/airways/mediastinum.
10. Severe cardiovascular disease:

    * Significant arrhythmias (requiring intervention), QTcF ≥450 ms (M)/470 ms (F)
    * ACS/heart failure/stroke/TIA within 6 months
    * NYHA class ≥II or LVEF <50%
    * Uncontrolled hypertension (≥160/100 mmHg despite ≥2 agents).
11. Abdominal fistula/GI perforation/abscess within 6 months.
12. Bowel obstruction/clinical signs of GI obstruction within 6 months.
13. Non-healing wounds, active ulcers, or untreated fractures.
14. Active autoimmune diseases or history of autoimmune diseases with potential recurrence (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism [patients with hypothyroidism controlled by hormone replacement therapy alone are not excluded]). Note: Patients with non-systemic skin conditions (e.g., vitiligo, psoriasis, alopecia), well-controlled type 1 diabetes on insulin, or childhood asthma with complete remission in adulthood requiring no intervention may be enrolled. Asthma patients requiring bronchodilator therapy are excluded.
15. Immunosuppressants (>10 mg/day prednisone equivalent) within 2 weeks.
16. Severe hypersensitivity to monoclonal antibodies.
17. Hepatic encephalopathy or CNS metastases.
18. Organ transplant history.
19. Symptomatic ascites requiring drainage within 3 months.
20. Uncontrolled hypertension (≥140/90 mmHg despite treatment).
21. Arterial/venous thrombosis within 6 months (stroke, DVT, PE).
22. Bleeding/thrombotic disorders (hemophilia, coagulopathy, thrombocytopenia).
23. Proteinuria ≥++ with 24-h urine protein >1.0 g.
24. Active infection (fever ≥38.5°C within 7 days or WBC >15×10⁹/L).
25. Interstitial lung disease (current or steroid-requiring history).
26. Active tuberculosis (confirmed by imaging/sputum/clinical assessment).
27. Immunodeficiency (HIV/syphilis).
28. Severe infection within 4 weeks (hospitalization required) or antibiotics within 2 weeks (prophylaxis allowed).
29. Recent treatments:

    * Liver surgery/HCC locoregional therapy within 4 weeks
    * Palliative bone radiotherapy within 2 weeks
    * Anti-HCC herbal medicine within 2 weeks
    * Unresolved toxicities (>Grade 1 per CTCAE v5.0, except alopecia).
30. Immunomodulators (interferons, interleukins) within 2 weeks.
31. Other investigational drugs within 4 weeks.
32. Allogeneic stem cell/organ transplant.
33. HBV-HCV coinfection.
34. Hypersensitivity to trial drug components/monoclonal antibodies/antiangiogenic agents.
35. Live vaccines within 4 weeks or planned during study.
36. Major surgery within 4 weeks or planned during study (biopsies/IV catheterization allowed).
37. Other exclusionary factors per investigator judgment (substance abuse, severe comorbidities, psychosocial risks).

Ages: 18 Days to 65 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 | From date of first dose of study drug until disease progression (up to approximately 3 years)
  ORR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by RECIST 1.1.

SECONDARY OUTCOMES:
Objective response rate (ORR) by mRECIST | From date of first dose of study drug until disease progression (up to approximately 3 years)
  ORR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by mRECIST.
The disease control rate (DCR) | From date of first dose of study drug until disease progression, stable disease (up to approximately 3 years)
  DCR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) or stable disease (SD) at the time of data cutoff as assessed by RECIST 1.1 and mRECIST.
The time to response (TTR) | From date of first dose of study drug to the date of first documentation of CR or PR (up to approximately 3 years)
  TTR was calculated as the time from treatment initiation to first documented response as assessed by RECIST 1.1 and mRECIST.
Duration of response (DOR) by RECIST 1.1 and mRECIST | From the first documentation of CR or PR to the first date of documentation of disease progression or death whichever occurs first (up to approximately 3 years)
  DOR is defined as the time from the first documentation of CR or PR to the date of first documentation of disease progression as assessed by RECIST 1.1 and mRECIST or death (whichever occurs first).
The progression-free survival time (PFS) | From date of first dose of study drug to the date of first documentation of disease progression or death (up to approximately 3 years)
  The progression-free survival time (PFS) defined as the time from the first study dose date to the date of first documentation of disease progression as assessed by RECIST 1.1 and mRECIST or death, whichever comes earlier.
The median overall survival time (OS) | From the start date of the Treatment Phase until date of death from any cause (up to approximately 3 years)
  OS is measured from the start date of the Treatment Phase (date of first study dose) until date of death from any cause. Participants who are lost to follow-up and the participants who are alive at the date of data cutoff will be censored at the date the participant was last known alive or the cut-off date.
The progression-free survival rate (PFSR) by RECIST 1.1 and mRECIST | From date of first dose of study drug to the date of first documentation of disease progression or death, whichever occurs first (up to approximately 3 years)
The overall survival rate (OSR) | From date of first dose of study drug to the date of documentation of death from any cause (up to approximately 3 years)
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | From the start date of the Treatment Phase until date of death from any cause (up to approximately 3 years)
Exploratory outcome measure: The quality of life (QoL) | From date of first dose of study drug to the date of first documentation of disease progression within the liver or death (up to approximately 3 years)
  The exploratory endpoint was the QoL, which was assessed using the European Organisation for Research and Treatment of Cancer QoL questionnaire (EORTC QLQ-C30).

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Hong Wu, Professor, Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan (SAP), and Clinical Study Report (CSR)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 3 months and ending 1 years after the publication of results.
Access Criteria: Data will be shared with qualified researchers who:
  1. Submit a scientifically valid research proposal with defined objectives and statistical analysis plans
  2. Require individual participant data (IPD) to address research questions not covered in the original publication
  3. Provide institutional ethics approval for the proposed secondary analysis
  4. Sign a Data Use Agreement (DUA) committing to:
     * Protect participant confidentiality
     * Not attempt to re-identify participants
     * Not transfer data to third parties
     * Destroy data after analysis completion